CLINICAL TRIAL: NCT05266716
Title: Field Study of a Digital Therapeutic Platform to Facilitate Treatment for Methamphetamine-Primary Stimulant Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affect Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Methamphetamine Field Study
Record Dates: First submitted 2022-01-07; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Methamphetamine Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Arm (Experimental): The study will involve a total of approximately 48 individuals enrolled during a six-week period as participants in the field test of the Affect digital therapeutic platform
  Interventions: Behavioral: Affect Methamphetamine Treatment Program

INTERVENTIONS:
Behavioral: Affect Methamphetamine Treatment Program — Components of the treatment services include: contingency management (CM; monetary incentives for drug tests negative for stimulants), the digital behavioral therapy curriculum (based on CBT) delivered via the Affect app on smartphones, weekly one-on-one telemedicine (TM) with clinical personnel and group therapy, and referral to psychiatrist for medication support, as needed. The program incrementally builds skills and beliefs to develop personally meaningful strategies to combat cravings, using such techniques as regular app-promoted deep breathing exercises, daily exercise, and help in making and sticking to a relapse prevention plan. Counseling sessions are arranged via text sent by the Team Care advocate and also presented to the participant via the app as a reminder. Individual and group therapy sessions occur over Zoom, which is integrated into the app.
  Contingency Management (CM). CM utilizes monetary incentives and rewards to promote behavior change.

SUMMARY:
The overall purpose of the observational, investigational pilot study is to assess the clinical utility of the Affect digital health platform (the Affect® "app") as part of the Affect program of treatment for methamphetamine-primary stimulant use disorder. The study also will identify elements of the Affect app that enhance engagement of participants in the study toward the goal of improving patient outcomes, including reduction/cessation of stimulant use.

DETAILED DESCRIPTION:
The research project is a single-group observational demonstration study to assess the clinical utility of a digital therapeutic technology (the Affect app) in terms of participant acceptance and the app's ability to enhance retention in the Affect program of services for the treatment of individuals with meth-primary stimulant use disorder (MUD). Measures of reduction and/or cessation of methamphetamine use will be assessed by saliva drug tests at least twice weekly during each participant's 8-week involvement in the program, at end of treatment, and via self-report at follow-up points at 1, 3, and 6 months after completion of the program. The app-based program will involve the same services for study participants as would occur regardless of the research, being a standard of care for MUD. The intervention phase of the study will be completed within approximately four months, with follow-ups of the final participants occurring approximately six months after the end of the intervention phase.

ELIGIBILITY:
To be eligible to participate in the study, prospective participants must:

1. Be 18 years of age or older;
2. Have methamphetamine use disorder (MUD) or documented high-risk methamphetamine use history, confirmed by DSM-5 criteria for stimulant use disorder, methamphetamine type;
3. Have stated interest in reducing and/or stopping methamphetamine use;
4. Have and be able to use a smartphone and agree to download and use the Affect app as part of treatment and study-related procedures;
5. Have a health insurance plan (or Medicaid) to ensure that participants have access to medical care if needed;
6. Be English speaking and have reading capacity sufficient to understand explanations of study procedures and the informed consent to participate;
7. Be a California resident with a mailing address or P.O. Box
8. Be able to freely give informed consent and be willing to electronically sign the digital informed consent to participate in the study;
9. Be willing to comply with study procedures, including use of the Affect app consistent with the study protocol and therapeutic activities.

III.6 EXCLUSION CRITERIA

Individuals will be precluded from enrolling in the study if they endorse (or if there is documentation of) any of following conditions. Already enrolled participants will be withdrawn from study participation upon emergence of any excluded condition (except pregnancy):

1. Serious medical diagnoses (e.g., seizure, stroke, heart disease);
2. Serious mental illness (e.g., schizophrenia, bipolar, active suicidality);
3. Moderate- to severe-level opioid use disorder or alcohol use disorder;
4. Pregnancy;
5. Have been in a prior study of pharmacological or behavioral treatment for MUD within 6 months of study consent;
6. Be concurrently receiving other behavioral or pharmacological services for treatment of MUD;
7. Have pending legal action or other situation that could inhibit consistent participation in the study or in study activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Participant retention in treatment | Up to 8 weeks through the duration of treatment
  Consistent with general approaches to measure retention (Hser et al., 2004, McLellan et al., 2006), the outcome will be based on completion as a binary measure at the end of the planned 8-week intervention for each participant. At the end-of-program telephone interview, participants will be deemed to be either treatment completers (i.e., retained) or dropouts (not retained if out of program before the end of week 4). Termination, expulsion, or unexplained non-response to or no contact with Affect personnel for more than seven consecutive days in any period of the 8-week study period equates to "drop-out" for the purpose of determining retention.
Participant participation in program | Up to 8 weeks through the duration of treatment
  The nature/degree of participation in this study is a construct composed of the number of successfully "attended" therapeutic tasks/events/activities per the Affect app relative to not-attended events such as: scheduled/planned digital/virtual interactions for program activities (e.g., counseling, group meetings), completed biological assessments (remote drug saliva tests), and kept appointments with referred service providers (e.g., psychiatrists, physicians).
Participant engagement with the Affect app | Up to 8 weeks through the duration of treatment
  Engagement with the Affect app components will be assessed via app-derived data on activity (i.e., duration, frequency, and consistency of involvement with app-directed tasks).
Participant satisfaction with the Affect app | Up to 8 weeks through the duration of treatment
  The investigators will assess the results of surveys/questionnaires/focus groups to characterize participant satisfaction with the app and importance of its features in the overall treatment program.
Effectiveness in reducing meth use | Up to 8 weeks through the duration of treatment
  The effectiveness measure is a composite of self-reported meth use (daily Yes/No) and meth-negative saliva test results (conducted remotely) over the course of each participant's 8-week duration in the program. A participant who provides at least 6 of 8 meth-negative saliva tests during the final 4 weeks of the 8-week program meets criteria for reduction/cessation of meth and thus demonstrates within-participant effectiveness of the program. Characteristics of the participants will be explored for possible associated factors that correlate with variations in outcomes across the sample.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zito, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Affect Therapeutics, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No participant data will be shared.

DOCUMENTS (1):
  • Informed Consent Form (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT05266716/ICF_000.pdf